CLINICAL TRIAL: NCT00977665
Title: A Multi-centered, Randomized, Double-blind, Placebo-controlled Clinical Trial to Assess the Efficacy, Safety, and Tolerability of Rasagiline Mesylate 1 mg in Patients With Multiple System Atrophy of the Parkinsonian Subtype (MSA-P)
Brief Title: Clinical Trial to Assess Efficacy, Safety, and Tolerability of Rasagiline Mesylate 1 mg in Patients With Multiple System Atrophy of the Parkinsonian Subtype (MSA-P)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Collaborators: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MSA-RAS-202; 2009-014644-11 (EudraCT Number)
Record Dates: First submitted 2009-09-15; First posted 2009-09-16 (Estimated); Results first posted 2015-02-26 (Estimated); Last update posted 2015-02-26 (Estimated); Status verified 2015-02

CONDITIONS: Multiple System Atrophy
MeSH Terms: conditions — Multiple System Atrophy | interventions — rasagiline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- rasagiline mesylate (Experimental): rasagiline tablet, 1 mg/day for up to 48 weeks.
  Interventions: Drug: rasagiline mesylate
- placebo (Placebo Comparator): placebo tablet for up to 48 weeks.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: rasagiline mesylate — rasagiline 1 mg tablet/day for 48 weeks
  Other Names: Azilect; TVP-1012
  Arms: rasagiline mesylate
Drug: placebo — placebo tablet for 48 weeks
  Arms: placebo

SUMMARY:
To test the clinical effect of rasagiline on subjects with MSA of the parkinsonian subtype.

ELIGIBILITY:
Inclusion Criteria:

* Subjects over 30 years old with a diagnosis of Possible or Probable MSA of the parkinsonian subtype (MSA-P) according to The Gilman Criteria (2008).
* Subjects who are less than 3 years from the time of documented MSA diagnosis.
* Subjects with an anticipated survival of at least 3 years in the opinion of the investigator.
* Subjects who are willing and able to give informed consent. Subjects who are not able to write may give verbal consent in the presence of at least one witness, and the witness should sign the informed consent form.

Exclusion Criteria:

* Subjects receiving treatment with midodrine or other sympathomimetics within 4 weeks prior to baseline visit.
* Subjects with severe orthostatic symptoms as assessed by a score of ≥ 3 on Unified Multiple System Atrophy Rating Scale (UMSARS) question 9.
* Subjects who meet any of the following criteria which tend to suggest advanced disease:

  1. Speech impairment as assessed by a score of ≥ 3 on UMSARS question 1
  2. Swallowing impairment as assessed by a score of ≥ 3 on UMSARS question 2
  3. Impairment in ambulation as assessed by a score of ≥ 3 on UMSARS question 7
  4. Falling more frequently than once per week as assessed by a score of ≥ 3 on UMSARS question 8
* Subjects taking disallowed medications according to the locally approved Azilect® label.
* Subjects taking monoamine oxidase (MAO) inhibitors within 3 months prior to baseline visit.
* Subjects with hypertension whose blood pressure, in the investigator's opinion, is not well controlled.
* Subjects who, based on the investigator's judgment, have a clinically significant or unstable medical or surgical condition that may preclude safe and complete study participation. Subjects with moderate or severe hepatic impairment.
* Subjects who have taken any investigational products within 60 days prior to baseline.
* Women of child-bearing potential who do not practice an acceptable method of birth control [acceptable methods of birth control in this study are: surgical sterilization, intrauterine devices, oral contraceptive, contraceptive patch, long-acting injectable contraceptive, partner's vasectomy, a double-protection method (condom or diaphragm with spermicide)].
* Pregnant or nursing women.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2009-12; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Werner Poewe, Prof, Principal Investigator — Innsbruck Medical University, Innsbruck, Austria
Locations (47):
- United States (15):
  - Teva Investigational Site 1004, Irvine, California
  - Teva Investigational Site 1014, La Jolla, California
  - Teva Investigational Site 1006, Sunnyvale, California
  - Teva Investigational Site 1010, Washington D.C., District of Columbia
  - Teva Investigational Site 1061, Boca Raton, Florida
  - Teva Investigational Site 1012, Tampa, Florida
  - Teva Investigational Site 1009, Worcester, Massachusetts
  - Teva Investigational Site 1003, Ann Arbor, Michigan
  - Teva Investigational Site 1007, Rochester, Minnesota
  - Teva Investigational Site 1011, St Louis, Missouri
  - Teva Investigational Site 1008, Rochester, New York
  - Teva Investigational Site 1001, Cleveland, Ohio
  - Teva Investigational Site 1002, Philadelphia, Pennsylvania
  - Teva Investigational Site 1013, Nashville, Tennessee
  - Teva Investigational Site 1005, Houston, Texas
- Austria (2):
  - Teva Investigational Site 3305, Graz
  - Teva Investigational Site 3304, Innsbruck
- Canada (4):
  - Teva Investigational Site 1109, Ottawa, Ontario
  - Teva Investigational Site 1111, Greenfield Park, Quebec
  - Teva Investigational Site 1108, Montreal, Quebec
  - Teva Investigational Site 1110, Québec, Quebec
- France (2):
  - Teva Investigational Site 3503, Lille
  - Teva Investigational Site 3502, Pessac
- Germany (6):
  - Teva Investigational Site 3206, Dresden
  - Teva Investigational Site 3203, Kiel
  - Teva Investigational Site 3201, Marburg
  - Teva Investigational Site 3205, München
  - Teva Investigational Site 3204, Tübingen
  - Teva Investigational Site 3202, Ulm
- Hungary (3):
  - Teva Investigational Site 5101, Budapest
  - Teva Investigational Site 5102, Debrecen
  - Teva Investigational Site 5103, Miskolc
- Israel (3):
  - Teva Investigational Site 8002, Ramat Gan, IL
  - Teva Investigational Site 8004, Haifa
  - Teva Investigational Site 8003, Tel Aviv
- Italy (3):
  - Teva Investigational Site 3006, Bologna
  - Teva Investigational Site 3004, Roma
  - Teva Investigational Site 3005, Venezia - Lido
- Netherlands (2):
  - Teva Investigational Site 3801, Amersfoort
  - Teva Investigational Site 3802, Sittard-Geleen
- Teva Investigational Site 3603, Lisbon, Portugal
- Spain (3):
  - Teva Investigational Site 3101, Barcelona
  - Teva Investigational Site 3102, Barcelona
  - Teva Investigational Site 3103, Seville
- United Kingdom (3):
  - Teva Investigational Site 3403, Cardiff, Wales
  - Teva Investigational Site 3401, London
  - Teva Investigational Site 3402, Newcastle upon Tyne

REFERENCES:
- [Derived] Poewe W, Seppi K, Fitzer-Attas CJ, Wenning GK, Gilman S, Low PA, Giladi N, Barone P, Sampaio C, Eyal E, Rascol O; Rasagiline-for-MSA investigators. Efficacy of rasagiline in patients with the parkinsonian variant of multiple system atrophy: a randomised, placebo-controlled trial. Lancet Neurol. 2015 Feb;14(2):145-52. doi: 10.1016/S1474-4422(14)70288-1. Epub 2014 Dec 8. PMID 25498732

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Eligible participants were randomized in a 1:1 ratio to either active treatment or placebo.
Period: Overall Study
Arm/Group | Rasagiline Mesylate | Placebo
Started | 84 | 90
Completed | 63 | 75
Not Completed | 21 | 15
Not completed — Withdrawal by Subject | 1 | 3
Not completed — Physician Decision | 2 | 1
Not completed — Sponsor requested withdrawal | 0 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Death | 3 | 2
Not completed — Adverse Event | 14 | 7
Not completed — Treatment failure | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rasagiline Mesylate | Placebo | Total
Number analyzed (Participants) | 84 | 90 | 174
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.9 (8.5) | 65.1 (8.6) | 65.0 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 39 | 74
  Male | 49 | 51 | 100
Race/Ethnicity, Customized [Number; unit: participants]
  Asian/Oriental | 0 | 2 | 2
  Black of African Heritage | 2 | 0 | 2
  Black or African American | 0 | 2 | 2
  Caucasian | 81 | 85 | 166
  Unknown | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  Portugal | 2 | 3 | 5
  United States | 16 | 16 | 32
  France | 9 | 8 | 17
  Hungary | 11 | 10 | 21
  Canada | 10 | 10 | 20
  Spain | 4 | 3 | 7
  Austria | 3 | 4 | 7
  Israel | 9 | 12 | 21
  Germany | 7 | 12 | 19
  Netherlands | 3 | 2 | 5
  Italy | 8 | 8 | 16
  United Kingdom | 2 | 2 | 4
Weight [Mean (Standard Deviation); unit: kg] | 76.9 (15.9) | 76.8 (15.5) | 76.9 (15.6)
Height [Mean (Standard Deviation); unit: cm] | 168.0 (10.2) | 169.0 (8.9) | 168.5 (9.6)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 27.2 (4.4) | 26.8 (4.4) | 27.0 (4.4)
Multiple System Atrophy of the Parkinsonian Subtype (MSA-P) [Number; unit: participants] — Possible or Probable MSA of the parkinsonian subtype (MSA-P) is according to The Gilman Criteria (2008).
  * Possible MSA requires a sporadic, progressive adult-onset disease including parkinsonism and at least one feature suggesting autonomic dysfunction plus one other feature that may be a clinical or a neuroimaging abnormality.
  * Probable MSA requires a sporadic, progressive adult-onset disorder including rigorously defined autonomic failure and poorly levodopa-responsive parkinsonism.
  participants
    Possible MSA-P | 38 | 55 | 93
    Probable MSA-P | 46 | 35 | 81

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 48/Termination Visit in the Total Unified Multiple System Atrophy Rating Scale (UMSARS Part I and II)
Description: This outcome represents the sum of 2 UMSARS sub-scales: Part I: Historical Review that includes 12 items and Part II: Motor Examination that includes 14 items. All items range from 0 to 4. Each subscale score is the sum of its items and the total UMSARS score is the sum of all 26 items. Hence the total UMSARS score can range from 0 to 104, with 0 meaning no impairment and 104 indicating severe impairment. Negative change from baseline scores indicate improvement.
  In the case that 6 items or more (out of 26) were missing at a certain visit, the UMSARS score for that visit was assigned a missing value.
Time Frame: Day 0 (baseline), Week 48
Population: Modified Intention-To-Treat Analysis Set (mITT): all randomized participants who took at least one dose of the study drug and who had at least one post-baseline efficacy assessment were included in the principal efficacy analysis, according to the treatment group to which they were originally assigned.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Rasagiline Mesylate | Placebo
Number analyzed (Participants) | 81 | 90
units on a scale | 7.2 (1.186) | 7.8 (1.091)
Statistical Analysis 1: Comparison: Rasagiline Mesylate vs Placebo; Test type: Superiority or Other; p = 0.6984, repeated measures model — A priori threshold for statistical significance is 0.05; Fixed effects: categorical week in trial by treatment interaction, center, and baseline UMSARS score; Mean Difference (Final Values) = -0.603, 95% CI 2-sided [-3.677 to 2.470]

2. Secondary Outcome: Clinical Global Impression Improvement (CGI-I) at Week 48/Termination Visit
Description: Outcome measures the investigator's clinical impression of the participants' improvement at Week 48 as compared to Week 12. CGI scale range from 1-7, with 1=very much improved, 4= no change, and 7=very much worse.
  In order to maintain the overall (hypotheses about primary and key secondary endpoints) type I error at the 0.05 level an hierarchy will be employed as follows: If the primary endpoint will be found to be significant at a significance level of 0.05 then the first key secondary endpoint will be tested, if this endpoint will be found to be significant in a significance level of 0.05 then the second key secondary endpoint will be tested and so on. The 'key' secondary endpoints are outcomes 2-6.
Time Frame: Week 48
Population: Modified Intention-To-Treat Analysis Set (mITT): all randomized participants who took at least one dose of the study drug and who had at least one post-baseline efficacy assessment.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Rasagiline Mesylate | Placebo
Number analyzed (Participants) | 80 | 88
units on a scale | 4.9 (0.152) | 4.8 (0.139)

3. Secondary Outcome: Change From Baseline to Week 24 in Total Unified Multiple System Atrophy Rating Scale (UMSARS) Score
Description: The UMSARS is composed of 2 sub-scales: Part I: Historical Review that includes 12 items and Part II: Motor Examination that includes 14 items. All items range from 0 to 4. Each subscale score is the sum of its items and the total UMSARS score is the sum of all 26 items. Hence the total UMSARS score can range from 0 to 104, with 0 meaning no impairment and 104 indicating severe impairment. Negative change from baseline scores indicate improvement.
  In the case that 6 items or more (out of 26) were missing at a certain visit, the UMSARS score for that visit was assigned a missing value.
Time Frame: Day 0 (baseline), Week 24
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Rasagiline Mesylate | Placebo
Number analyzed (Participants) | 81 | 90
units on a scale | 3.8 (0.811) | 3.0 (0.760)

4. Secondary Outcome: Percentage of Participants Who Achieved a Score of >=3 on the Unified Multiple System Atrophy Rating Scale (UMSARS) Question #7 Regarding Ambulation
Description: UMSARS' Question #7 concerns the participant's ability to walk, rated on a scale of 0=normal to 4=cannot walk at all even with assistance. This endpoint counts participants rated a 3 or worse. Rating 3 = Severely impaired; assistance and/or walking aid needed occasionally.
Time Frame: up to week 48
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Rasagiline Mesylate | Placebo
Number analyzed (Participants) | 81 | 90
percentage of participants | 46.4 | 52.2

5. Secondary Outcome: Mean Score of the Composite Autonomic Symptom Scale Select (COMPASS_Select Change) at Week 48/Termination Visit
Description: COMPASS_Select change is comprised of 5 of the 11 domains in the COMPASS scale: Orthostatic Intolerance, Bladder Disorder, Sweating, Vasomotor, and Sleep Disorder COMPASS_Select change has a range of -150 to 150, with -150 indicating symptoms are much better and 150 indicating symptoms are much worse.
Time Frame: 48 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Rasagiline Mesylate | Placebo
Number analyzed (Participants) | 79 | 90
units on a scale | 34.1 (4.342) | 42.7 (4.025)

6. Secondary Outcome: Change From Baseline to Week 48/Termination Visit in the Multiple System Atrophy (MSA) Health-related Quality of Life (QoL) Scale
Description: The Multiple System Atrophy Quality of Life questionnaire (MSA-QoL) is a self-reported questionnaire focusing on MSA-specific symptoms and has a scale ranging from 0 - 160, with 0= 'no problem' and 160= "extreme problem".
Time Frame: Day 0 (baseline), Week 48
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Rasagiline Mesylate | Placebo
Number analyzed (Participants) | 74 | 82
units on a scale | 4.6 (2.877) | 9.3 (2.720)

7. Secondary Outcome: Rate of Progression in Total Unified Multiple System Atrophy Rating Scale (UMSARS) Score From Baseline to Weeks 12-48
Description: The UMSARS is composed of 2 sub-scales: Part I: Historical Review that includes 12 items and Part II: Motor Examination that includes 14 items. All items range from 0 to 4. Each subscale score is the sum of its items and the total UMSARS score is the sum of all 26 items. Hence the total UMSARS score can range from 0 to 104, with 0 meaning no impairment and 104 indicating severe impairment.
  The rate of progression of atrophy is represented by the slope of change from baseline scores for visits between Weeks 12 and 48.
Time Frame: Day 0 (baseline), Weeks 12-48
Population: as for outcome 2
Measure: Mean (Standard Error); unit: units on a scale/week
Arm/Group | Rasagiline Mesylate | Placebo
Number analyzed (Participants) | 81 | 90
units on a scale/week | 0.1496 (0.02843) | 0.1788 (0.02591)

8. Secondary Outcome: Change From Baseline to Week 48 or Termination in UMSARS Subscores for Parts I, II and IV
Description: UMSARS Part I is an historical review and scores symptoms of neurological and autonomic dysfunction with 12 items rated on a scale of 0 (normal) to 4 (extreme dysfunction). The full scale for Part 1 is therefore 0 (normal) to 48 (extreme dysfunction). Part II is a motor examination and has 14 items also rated on a scale of 0 to 4 for a full scale of 0 (normal) to 56 (extreme dysfunction). Part IV is a global disability scale with rates the extent of disease from 1 (normal) to 5 (severe disease).
Time Frame: Day 0 (baseline), Week 48 or termination visit
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Rasagiline Mesylate | Placebo
Number analyzed (Participants) | 81 | 90
units on a scale
  UMSARS Part I | 3.8233 (0.6339) | 4.3785 (0.5808)
  UMSARS Part II | 3.6478 (0.7017) | 3.5068 (0.6445)
  UMSARS Part IV | 0.7100 (0.1040) | 0.6763 (0.09523)

9. Secondary Outcome: Change From Baseline to Week 12 in Total UMSARS Score for Symptomatic Effect
Description: This outcome represents the sum of 2 UMSARS sub-scales: Part I: Historical Review that includes 12 items and Part II: Motor Examination that includes 14 items. All items range from 0 to 4. Each subscale score is the sum of its items and the total UMSARS score is the sum of all 26 items. Hence the total UMSARS score can range from 0 to 104, with 0 meaning no impairment and 104 indicating severe impairment. Negative change from baseline scores indicate improvement.
Time Frame: Day 0 (baseline), Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rasagiline Mesylate | Placebo
Number analyzed (Participants) | 79 | 88
units on a scale | 1.875 (0.693) | 1.574 (0.678)

10. Secondary Outcome: Estimates for Time to Change in Anti-Parkinsonian or Anti-Orthostatis Hypotension Medications
Description: Change in anti-parkinsonian or anti-orthostatic hypotension medication is defined by at least one of the following events:
  1. An addition of a new anti-parkinsonian or anti-orthostatic hypotension medication during study.
  2. Dose modification of anti-parkinsonian or anti-orthostatic hypotension concomitant medications reflecting disease progression.
  The event of interest, determined on a by patient basis, therefore, is the earliest event of the two events defined above. Otherwise, patient is right censored according to his/her study termination date.
  Since less than 25% of participants had an event, median estimatation for time to change in medications is not possible.
Time Frame: Day 0 (baseline) to Week 48 or termination visit
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Rasagiline Mesylate | Placebo
Number analyzed (Participants) | 84 | 90
days | 246 [162 to NA] — Not enough participants had an event for which to a median or upper 95% CI for the 25th percentile can be estimated, hence only the 25th percentile estimate and the lower 95% CI for the 25th percentile are presented | 294 [226 to NA] — Not enough participants had an event for which to a median or upper 95% CI for the 25th percentile can be estimated, hence only the 25th percentile estimate and the lower 95% CI for the 25th percentile are presented
Statistical Analysis 1: Comparison: Rasagiline Mesylate vs Placebo; Test type: Superiority or Other; Hazard Ratio (HR) = 1.189, 95% CI 2-sided [0.646 to 2.186]

11. Secondary Outcome: Change From Baseline to Week 48 or Termination in the Montreal Cognitive Assessment Scale (MoCA) Scale
Description: MoCA is a cognitive screening test which helps health professionals identify mild cognitive impairment. The total scale is 0 (significant cognitive impairment) to 30 (no impairment detected). Scores >=26 are considered normal. Positive change from baseline scores indicate improvement in cognition.
Time Frame: Day 0 (baseline), Week 48 or termination visit
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Rasagiline Mesylate | Placebo
Number analyzed (Participants) | 73 | 82
units on a scale | -1.1572 (0.4590) | -0.5786 (0.4186)

12. Secondary Outcome: Percentage of Participants Who Achieved a Score of >=3 on the Unified Multiple System Atrophy Rating Scale (UMSARS) Question #1 (Speech Impairment), Question #2 (Swallowing Impairment) and Question #8 (Falling)
Description: UMSARS' questions are rated on a scale of 0=normal to 4=extreme impairment.
  This endpoint reports the percentage of participants rated a 3 or worse. Rating 3 = Severely impaired speech (Question #1), swallowing (Question #2) or falling more frequently than once per week (Question #8).
Time Frame: up to week 48
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Rasagiline Mesylate | Placebo
Number analyzed (Participants) | 81 | 90
percentage of participants
  Q1. Speech Impairment | 35.7 | 30.0
  Q2. Swallowing Impairment | 3.6 | 6.7
  Q8. Falling | 19.0 | 15.6

13. Secondary Outcome: Change From Baseline to Week 48 or Termination in the Beck Depression Inventory Scale (BDI-II)
Description: The Beck Depression Inventory (BDI-II), is a 21-question multiple-choice self-report inventory, one of the most widely used instruments for measuring the severity of depression. Participants are asked to pick the answer for each question that best describes the way they have been feeling in the past two weeks, including the day participants complete the questionnaire. Each question is rated on a scale of 0-3, with 0 meaning the participant does not feel the emotion described in the question, and 3 meaning the participant has extremely strong feelings. Total scale is 0 (no evidence of depression) to 63 (extreme depression). Negative change from baseline scores indicate improvement in level of depression.
Time Frame: Day 0 (baseline), Week 48 or termination visit
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Rasagiline Mesylate | Placebo
Number analyzed (Participants) | 72 | 82
units on a scale | 0.4894 (0.9988) | 0.7145 (0.9241)

14. Secondary Outcome: Total Number of Falls During the Study
Description: Participants recorded each time they fell during the study in a diary.
Time Frame: Day 1 up to week 48
Population: Modified Intention-To-Treat Analysis Set (mITT): all randomized participants who took at least one dose of the study drug and who had at least one post-baseline efficacy assessment, and who maintained diaries.
Measure: Median (Inter-Quartile Range); unit: falls
Arm/Group | Rasagiline Mesylate | Placebo
Number analyzed (Participants) | 79 | 89
falls | 4.00 [1.00 to 14.00] | 5.00 [1.00 to 10.00]

ADVERSE EVENTS:
Time Frame: Day 1 to Week 48
Arm/Group | Placebo | Rasagiline Mesylate
Serious Adverse Events (participants affected / at risk) | 23/90 | 29/84
Other Adverse Events (participants affected / at risk) | 45/90 | 41/84
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=90) | Rasagiline Mesylate (N=84)
ANAEMIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
CARDIAC FAILURE (Cardiac disorders) | 1 (1) | 0 (0)
CARDIOVASCULAR INSUFFICIENCY (Cardiac disorders) | 0 (0) | 1 (1)
CORONARY ARTERY DISEASE (Cardiac disorders) | 1 (1) | 0 (0)
LEFT VENTRICULAR FAILURE (Cardiac disorders) | 1 (1) | 0 (0)
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 0 (0) | 1 (1)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 1 (1) | 0 (0)
ABDOMINAL RIGIDITY (Gastrointestinal disorders) | 0 (0) | 1 (1)
ACUTE ABDOMEN (Gastrointestinal disorders) | 0 (0) | 1 (1)
CONSTIPATION (Gastrointestinal disorders) | 1 (1) | 1 (1)
CROHN'S DISEASE (Gastrointestinal disorders) | 0 (0) | 1 (1)
GASTRIC ULCER (Gastrointestinal disorders) | 1 (1) | 0 (0)
HAEMATEMESIS (Gastrointestinal disorders) | 0 (0) | 1 (1)
ASTHENIA (General disorders) | 1 (1) | 0 (0)
CHEST PAIN (General disorders) | 0 (0) | 1 (1)
CHILLS (General disorders) | 1 (1) | 0 (0)
FATIGUE (General disorders) | 1 (1) | 0 (0)
OEDEMA PERIPHERAL (General disorders) | 1 (1) | 0 (0)
PYREXIA (General disorders) | 1 (1) | 1 (2)
CHOLECYSTITIS (Hepatobiliary disorders) | 1 (1) | 0 (0)
ARTHRITIS INFECTIVE (Infections and infestations) | 0 (0) | 1 (1)
CARBUNCLE (Infections and infestations) | 0 (0) | 1 (1)
CYSTITIS (Infections and infestations) | 0 (0) | 1 (1)
DEVICE RELATED INFECTION (Infections and infestations) | 1 (1) | 0 (0)
HERPES ZOSTER (Infections and infestations) | 1 (1) | 0 (0)
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (1)
LUNG INFECTION (Infections and infestations) | 0 (0) | 1 (1)
NASOPHARYNGITIS (Infections and infestations) | 0 (0) | 1 (1)
PNEUMONIA (Infections and infestations) | 1 (1) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 1 (1) | 4 (6)
FALL (Injury, poisoning and procedural complications) | 3 (3) | 2 (2)
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
HEAD INJURY (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
HIP FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
LACERATION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
LUMBAR VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
PUBIS FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
WEIGHT DECREASED (Investigations) | 1 (1) | 0 (0)
DECREASED APPETITE (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
HEADACHE (Nervous system disorders) | 1 (1) | 0 (0)
HYPOKINESIA (Nervous system disorders) | 1 (1) | 0 (0)
LOSS OF CONSCIOUSNESS (Nervous system disorders) | 0 (0) | 1 (1)
SYNCOPE (Nervous system disorders) | 2 (2) | 2 (2)
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 0 (0) | 1 (1)
DELIRIUM (Psychiatric disorders) | 0 (0) | 1 (1)
MENTAL STATUS CHANGES (Psychiatric disorders) | 1 (1) | 0 (0)
SLEEP DISORDER (Psychiatric disorders) | 1 (1) | 0 (0)
SUICIDE ATTEMPT (Psychiatric disorders) | 1 (1) | 0 (0)
HAEMATURIA (Renal and urinary disorders) | 1 (1) | 0 (0)
URINARY RETENTION (Renal and urinary disorders) | 1 (1) | 1 (1)
URINARY TRACT OBSTRUCTION (Renal and urinary disorders) | 1 (1) | 0 (0)
BENIGN PROSTATIC HYPERPLASIA (Reproductive system and breast disorders) | 1 (1) | 1 (1)
PROSTATOMEGALY (Reproductive system and breast disorders) | 0 (0) | 1 (1)
CHOKING (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
DYSPHONIA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (3)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
RESPIRATORY DISTRESS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
CATARACT OPERATION (Surgical and medical procedures) | 1 (2) | 0 (0)
GASTROSTOMY (Surgical and medical procedures) | 0 (0) | 1 (1)
HIP ARTHROPLASTY (Surgical and medical procedures) | 0 (0) | 1 (1)
INGUINAL HERNIA REPAIR (Surgical and medical procedures) | 0 (0) | 1 (1)
KNEE ARTHROPLASTY (Surgical and medical procedures) | 0 (0) | 1 (1)
PROSTATECTOMY (Surgical and medical procedures) | 0 (0) | 1 (1)
TRACHEOSTOMY (Surgical and medical procedures) | 0 (0) | 1 (1)
TRANSURETHRAL PROSTATECTOMY (Surgical and medical procedures) | 0 (0) | 1 (1)
HYPERTENSION (Vascular disorders) | 1 (1) | 0 (0)
LABILE BLOOD PRESSURE (Vascular disorders) | 0 (0) | 1 (1)
ORTHOSTATIC HYPOTENSION (Vascular disorders) | 0 (0) | 3 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=90) | Rasagiline Mesylate (N=84)
CONSTIPATION (Gastrointestinal disorders) | 5 (6) | 5 (5)
OEDEMA PERIPHERAL (General disorders) | 6 (6) | 9 (9)
NASOPHARYNGITIS (Infections and infestations) | 6 (6) | 4 (4)
URINARY TRACT INFECTION (Infections and infestations) | 12 (22) | 6 (14)
FALL (Injury, poisoning and procedural complications) | 9 (12) | 5 (6)
DIZZINESS (Nervous system disorders) | 10 (14) | 10 (11)
HEADACHE (Nervous system disorders) | 7 (7) | 3 (3)
SOMNOLENCE (Nervous system disorders) | 5 (6) | 2 (2)
DEPRESSION (Psychiatric disorders) | 5 (5) | 1 (1)
ORTHOSTATIC HYPOTENSION (Vascular disorders) | 3 (3) | 6 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.